CLINICAL TRIAL: NCT01701960
Title: Effect of Local Anesthetic on Hemodynamic Measures During Nasal Surgery
Status: Withdrawn | Type: Observational
Why Stopped: no time
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kristin Seiberling, MD, Associate Professor, Loma Linda University
Other Study IDs: 5120227
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Heart Rate; Blood Pressure; Blood Loss During Surgery; Surgical Field

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: This cohort will be injected with 1% lidocaine with 1:100,000 of epinephrine into the nasal mucosa at the time of nasal surgery
- Group 2: This group will be injected with 1% lidocaine with 1:200,000 of epinephrine into the nasal mucosa at the start of nasal surgery.

SUMMARY:
1% Lidocaine with 1:100,000 to 1:200,000 of epinephrine is routinely injected into the nasal mucosa during nasal surgery to reduce patient blood loss and improve the surgical field and visibility. Typically 1% lidocaine with 1:100,000 of epinephrine is used in nasal surgery. However, 1 % lidocaine with 1:200,000 (which is a more dilute solution of epinephrine) is also used. This latter dose theoretically should have a lesser effect on cardiac stimulation which increases the heart rate and blood pressure at the time of surgery. The nasal mucosa has excellent absorbing ability which is great for the application of drugs but there is concern for systemic absorption and side effects. Potential serious side effects can occur with local injection such as hypertension, tachycardia, and cardiac arrhythmias. These side effects occur mainly through the absorption of epinephrine. It is the goal of this study to see if a weaker concentration of epinephrine (1:200,000) can maintain a good surgical field with a decrease in hemodynamic side effects.

DETAILED DESCRIPTION:
Objective- To evaluate the effect of 1% lidocaine with 1:200,000 of epinephrine on hemodynamic measures and bleeding in the surgical field in patients undergoing nasal surgery compared to 1% lidocaine with 1:100,000.

Recruitment plan- Patients undergoing general anesthetic for nasal surgery (septoplasty or sinus surgery) will be asked to participate in this study. All patients undergoing nasal surgery are injected with local anesthetic into the nasal mucosa after induction of general anesthetic. Those patients who agree to participate in the study will be randomized into 2 groups (injection either 1 % lidocaine with 1:100,000 or 1:200,000 of epinephrine).

Procedures

1. Patients will be put to sleep following standard general anesthetic protocol
2. Patients will be injected with either 1% lidocaine with 1:100,000 or 1% lidocaine with 1:200,000 into the nasal mucosa
3. After injection the following will be measured every 15 minutes for the first hour to evaluate effectiveness of the local anesthetic.

   1. Heart rate
   2. Blood pressure
   3. Routine ECG monitoring
   4. MAP (mean arterial pressure)
   5. Surgical field, degree of bleeding.

Alternatives- Subjects can refuse to participate in the study. If subjects refuse to participate in the study they will still be injected with 1% lidocaine with 1:200,000 of epinephrine which is standard of care

Data analysis- data will be compiled and statistical analysis will be made using PRISM software.

ELIGIBILITY:
Inclusion Criteria:

* any patient between the ages of 16-75 who is scheduled to undergo routine nasal surgery.

Exclusion Criteria:

* allergy to lidocaine,
* recent MI,
* recent stroke,
* uncontrolled hypertension,
* arrhythmias,
* congestive heart failure.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects ages 16-75 undergoing routine nasal surgery which will include septoplasty and sinus surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change in blood pressure | over the course of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Seiberling, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States